CLINICAL TRIAL: NCT00857077
Title: Evaluation of the Safety and Effectiveness of EPI-linked Malaria Intermittent Chemotherapy and Iron Supplementation
Brief Title: Intermittent Preventive Treatment for Malaria in Infants in Navrongo Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Navrongo Health Research Centre, Navrongo, Ghana. (Unknown); Kintampo Health Research Centre, Ghana (Other); INDEPTH Network (Other); Department for International Development, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DFID-R7602
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Anaemia; Malaria
Keywords: incidence of anaemia
MeSH Terms: conditions — Anemia; Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 Sulfadoxine-pyrimethamine (SP) (Active Comparator)
  Interventions: Drug: Sulfadoxine-pyrimethamine

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine
  Arms: 2 Sulfadoxine-pyrimethamine (SP)
Drug: Placebo
  Arms: 1 Placebo

SUMMARY:
Evaluation of the safety and effectiveness of malaria intermittent chemotherapy and iron supplementation delivered through Expanded Programme on Immunisation vaccination clinics.

DETAILED DESCRIPTION:
Anaemia is one of the main disease burdens of children in developing countries. Severe anaemia is often fatal, while moderate anaemia leads to growth and cognitive disorders. The incidence of anaemia in children is extremely high in malaria endemic areas since episodes of clinical malaria and asymptomatic parasitaemia result in red cell destruction. It has been shown in Tanzania that the incidence of severe anaemia in infants can be reduced by 30% by regular administration of iron supplements, and by 60% if regular malaria chemoprophylaxis is given in addition. One way to operationalise this research finding, with minimal additional cost to governments and communities, is to link the distribution of iron and antimalarial drugs to the EPI programme. We propose a community-randomised trial to study the effectiveness of intermittent iron supplements and malaria chemotherapy in reducing the incidence of anaemia and clinical malaria, and to investigate any possible interactions of iron and antimalarial drugs with EPI vaccines. The study will have two arms: children in both arms will receive monthly supplies of twice weekly iron supplements when they attend EPI and growth monitoring clinics. In addition, children in arm 1 will receive a placebo when they receive Polio/DPT 2, Polio/DPT 3 and measles vaccines, while those in arm 2 will receive sulfadoxine-pyrimethamine (SP). The baseline incidence of anaemia and malaria, and immune response to EPI vaccines, will be estimated in a sample of children from a non-intervention area adjacent to the study area. The immune response to EPI vaccines, drug side-effects, and the incidence of anaemia and malaria will be compared between the two arms of the study and with the non-intervention area. Any possible 'rebound' in malaria incidence due to impairment of immunity will be monitored and treated during the six months after stopping the chemotherapy and supplementation.

ELIGIBILITY:
Inclusion Criteria:

* All infants living in study clusters without a history of allergy to sulfadoxine-pyrimethamine were eligible for enrollment in the study.

Exclusion Criteria:

* History of allergy to sulfadoxine-pyrimethamine.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2485 (Actual)
Dates: Start 2000-09; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
incidence of anaemia

SECONDARY OUTCOMES:
incidence of clinical malaria
incidence of severe disease and mortality
prevalence of anaemia and parasitaemia
incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chandramohan, MD; PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Brian Greenwood, MD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Navrongo Health Research Centre, Navrongo, Upper East Region, Ghana

REFERENCES:
- [Result] Chandramohan D, Owusu-Agyei S, Carneiro I, Awine T, Amponsa-Achiano K, Mensah N, Jaffar S, Baiden R, Hodgson A, Binka F, Greenwood B. Cluster randomised trial of intermittent preventive treatment for malaria in infants in area of high, seasonal transmission in Ghana. BMJ. 2005 Oct 1;331(7519):727-33. doi: 10.1136/bmj.331.7519.727. PMID 16195288